CLINICAL TRIAL: NCT01056874
Title: Open-Label, Fixed Sequence, Crossover Study To Estimate The Effect Of Multiple Dose Maraviroc On Single Dose Digoxin Pharmacokinetics In Healthy Subjects
Brief Title: Effect Of Maraviroc On The Pharmacokinetics Of Digoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A4001097
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Healthy; HIV Infections
Keywords: Maraviroc; Digoxin; P-glycoprotein; Pharmacokinetics; Drug Interaction; HIV
MeSH Terms: conditions — HIV Infections | interventions — Digoxin; Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Digoxin (Active Comparator)
  Interventions: Drug: Digoxin
- Digoxin + Maraviroc (Experimental)
  Interventions: Drug: Digoxin; Drug: Maraviroc

INTERVENTIONS:
Drug: Digoxin — Oral Digoxin 0.25 mg single dose
  Arms: Digoxin
Drug: Digoxin — Oral Digoxin 0.25 mg single dose on Day 5
  Arms: Digoxin + Maraviroc
Drug: Maraviroc — Oral Maraviroc 300 mg twice daily for 6 days
  Other Names: Selzentry, Celsentri
  Arms: Digoxin + Maraviroc

SUMMARY:
This is an open labelled study to estimate the effect of maraviroc on the pharmacokinetics of digoxin, a probe for p-glycoprotein.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 25.5 kg/m2.
* Total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
* Subjects with an estimated creatinine clearance (CLcr) <80 ml/min.
* Pregnant or nursing females.
* Females of childbearing potential who are unwilling or unable to use an acceptable method of contraception as outlined in this protocol from at least 14 days prior to the first dose of study medication until completion of study.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To estimate the effect of multiple dose maraviroc on the pharmacokinetics of digoxin. | 21 days

SECONDARY OUTCOMES:
To investigate the safety and tolerability of maraviroc and digoxin when co-administered. | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001097&StudyName=Effect%20Of%20Maraviroc%20On%20The%20Pharmacokinetics%20Of%20Digoxin